CLINICAL TRIAL: NCT01128140
Title: Motivating Treatment Seeking and Behavior Change by Untreated Military Personnel Abusing Alcohol or Drugs
Brief Title: Efficacy Trial of Warrior Check-Up
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Denise Walker, Research Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37278-C
Record Dates: First submitted 2010-05-14; First posted 2010-05-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Alcohol Abuse; Alcohol Dependence; Substance Abuse; Substance Dependence
Keywords: motivational enhancement therapy
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Motivational Interviewing; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Enhancement Therapy (Experimental)
  Interventions: Behavioral: Motivational Enhancement Therapy
- Education (Active Comparator)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — MET, a 30-60 minute telephone session, seeks to increase motivation for change by highlighting inconsistencies between substance use behaviors and beliefs and negative consequences experienced as a result of the behaviors. The counselor will guide the participant in reviewing the Personal Feedback Report (PFR), using MI strategies to elicit the participant's reactions and foster motivation for change. The PFR will show the participant's self-reported alcohol and drug use behavior, consequences of SA, and the participant's perceived and actual descriptive norms for SA behavior. The second phase will target strengthening commitment to change. Counselors will explore with participants the pros and cons of seeking treatment. As the participant verbalizes potential benefits of learning more about treatment, the counselor will use MI skills to encourage elaboration of his/her thinking with the goal of tipping the scale toward a decision to consider taking steps toward treatment.
  Arms: Motivational Enhancement Therapy
Behavioral: Education — Participants will receive educational information on the health, psychological, social, and legal consequences of substance abuse. Included in the session will be: legal and behavioral definitions of SA, the social and legal consequences of SA, impact of SA on military duty, a review of the policies on substance use in the military, and treatment resources. The session will be conducted via the telephone and will last from 30-60 minutes. Counselors will present information in a didactic manner and will avoid the use of Motivational Interviewing skills (reflective listening, developing discrepancy, reinforcing participant statements regarding change).
  Arms: Education

SUMMARY:
This study will develop and test a brief telephone-delivered motivational enhancement intervention for substance abusing military personnel who are not currently in treatment. The hypotheses being tested are that this intervention will prompt a willingness to participate voluntarily in a self-appraisal of substance abuse behavior and consequences, self-initiated change or enrollment in a treatment or self-help program, and cessation of abuse of alcohol or other drugs.

DETAILED DESCRIPTION:
The health and well-being of military personnel, and consequently the capacity for optimal functioning of military units, are compromised by the abuse of alcohol and/or other drugs. Rates of heavy drinking are higher among military personnel than in the general population and are even higher among recently deployed personnel.

While counseling can be effective, most substance abusers do not tend to voluntarily seek treatment. Moreover, military personnel encounter more real and perceived barriers to seeking treatment.

The substance abuse field is increasingly focusing on developing interventions for those at early stages of readiness to change, i.e., those contemplating but not yet committed to change. A brief, telephone-delivered motivational enhancement intervention (MET) called a "check-up," has shown promise in promoting self-initiated behavior change as well as voluntary treatment entry, enhanced retention, and more successful outcomes for substance abuse.

Adapting the "check-up" for application with military personnel is warranted for three key reasons: (1) it has the potential of overcoming barriers to treatment-seeking, i.e., stigma and apprehension of a negative impact on one's military career; (2) it has the potential of attracting voluntary participation; and (3) protocols for disseminating this low cost intervention for use with deployed military can readily be developed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. current abuse or dependence on one or more substances
2. not currently enrolled in a counseling program focusing on substance abuse
3. currently serving in the Army or other branch of the military.

Exclusion Criteria:

1. non-fluency in English
2. evidence of psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Form 90D | 3 months
  Structured interview that uses a timeline follow-back procedure to elicit detailed daily information on the use of alcohol and other drugs.
Inventory of Drug Use Consequences | 3 months
  A 50-item inventory of consequences related to alcohol and drug use.
Treatment Seeking and Preparation Behaviors Questionnaire | 3 months
  Assesses treatment-seeking attitudes, intentions, and behaviors.

SECONDARY OUTCOMES:
Stages of Change Readiness and Treatment Eagerness Scale | 3 months
  19-item questionnaire that assesses readiness to make changes in alcohol or drug use behaviors.
Drinking Norms Rating Form | 3 months
  Participant estimates of prevalence and frequency/volume of alcohol/drug consumption by the average person and the average person in the military.

CONTACTS AND LOCATIONS:
Overall Officials: Denise D Walker, PhD, Principal Investigator — University of Washington School of Social Work
Locations (1):
- University of Washington Innovative Programs Research Group, Seattle, Washington, United States

REFERENCES:
- [Derived] Rodriguez LM, Neighbors C, Walker D, Walton T. Mechanisms and moderators of intervention efficacy for soldiers with untreated alcohol use disorder. J Consult Clin Psychol. 2020 Feb;88(2):137-148. doi: 10.1037/ccp0000471. PMID 31894995